CLINICAL TRIAL: NCT06669130
Title: Efficacy and Safety of Xiangtong TM Full Degradation Sinus Drug Stent System
Brief Title: Xiangtong TM Full Degradation Sinus Drug Stent System Prospective, Open, Single-center, Randomized Controlled Clinical Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-SR-350
Record Dates: First submitted 2024-10-30; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Chronic Rhinosinusitis (CRS)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Xiangtong TM full degradation sinus drug stent system (Experimental)
  Interventions: Device: Xiangtong TM full degradation sinus drug stent system
- nasopore (Placebo Comparator)
  Interventions: Device: nasopore

INTERVENTIONS:
Device: Xiangtong TM full degradation sinus drug stent system — use Xiangtong TM full degradation sinus drug stent system to deliver drugs into sinus
  Arms: Xiangtong TM full degradation sinus drug stent system
Device: nasopore — use nasopore to protect the post-operative sinus
  Arms: nasopore

SUMMARY:
Xiangtong® Fully Degradable Sinus Drug Stent System is a high-tech medical device independently developed by Puyi Bio, specially designed for patients with chronic rhinosinusitis (CRS) undergoing endoscopic sinus surgery (ESS).The product is implanted into the target site during and after surgery, which not only supports the separation of the wound and fixes the repaired mucosal flap, but also controls edema, prevents adhesions, maintains smooth drainage, and sustains the target site to fight against inflammation and promotes healing by means of slow-release hormones.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are 18-65 years of age, male or non-pregnant female. The subject/legally authorized representative understands the purpose and procedures of the trial and voluntarily signs an informed consent form.

Subjects must meet the diagnostic guidelines for chronic rhinosinusitis, have a confirmed diagnosis of bilateral chronic rhinosinusitis, and have a CT scan confirming bilateral Lund-Mackay scores >6 (CT scan within 3 months prior to surgery is valid).

* Female subjects who are not breastfeeding at the time of the screening visit and who do not plan to breastfeed or become pregnant for up to one year after the starting point.
* Subject has not participated in another clinical trial in the previous 3 months and agrees not to participate in another clinical trial until the endpoints of this trial have been met.

Exclusion Criteria:

* Subject has a known allergic reaction or contraindication to the device material and its degradation products (mometasone acid, levulinic acid, racemic polylactic acid, propyl lactate, lactic acid).
* The subject is on long-term oral hormonal medications.
* The subject is receiving immunosuppressive therapy or has a known immunosuppressive or autoimmune disease: the subject has diabetes mellitus.
* The subject has or has had glaucoma or high intraocular pressure.
* The subject has cataracts.
* The subject has an artificial eye.
* Acute bacterial sinusitis and acute fungal sinusitis.
* Subject has a life expectancy of less than 12 months.
* Subject has participated in a clinical trial of another drug or device that did not meet the primary study endpoint: Subject is unable or unwilling to participate in this trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative reintervention rates based on imaging evaluations | 30 days after operation